CLINICAL TRIAL: NCT04286633
Title: The Influence of Lead and Cadmium Seminal Plasma Level on Intracytoplasmic Sperm Injection (ICSI) Outcome
Brief Title: Influence of Pb&Cd Seminal Plasma Level & ICSI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaimaa Mostafa Atef Abdul-Rahman, Doctor, Assiut University
Other Study IDs: Pb&Cd seminal level&ICSI
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Infertility, Male
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the influence of lead (pb) and cadmium (cd) seminal plasma level on embryo development and pregnancy rate during intracytoplasmic sperm injection (ICSI).

DETAILED DESCRIPTION:
The inability to have children, both by natural procreation and medically assisted reproduction, is not only a challenge for medical science but also an economic and social problem. Infertility is a complex disorder with multiple genetic and environmental causes (Gill et al.,2018) One of the factors that may be responsible for this phenomenon is contamination of the environment with heavy metals Two of the most widely-recognized reproductive toxins are lead (Pb) and cadmium (Cd) (Wdowiak et al., 2018).

Food, water and tobacco and smoking are the primary source of baseline exposure to lead and cadmium (Tong et al., 2000; Bernard, 2008) Each of cadmium and lead were inversely correlated with semen parameters as, ejaculate volume, sperm count, sperm concentration, live sperms and rapid mobility. ( Zaki et al.,2018).

Reproductive contaminants found in follicular fluid (FF) and seminal plasma may compromise the quality of oocytes and or sperm, which may become one of the risk factors for reproductive outcome. The data available suggests certain chemicals or their metabolite reaches the seminal plasma and/or FF, indicating their possible impact in In Vitro fertilization (IVF) outcome ,However, more studies are needed with regard to relationship between exposure level and affected parameters. (Kumar et al., 2010).

ELIGIBILITY:
Inclusion Criteria:

* Isolated male infertility (oligozoospermia, astenozoospermia, teratozoospermia)
* First ICSI cycle
* Female partner ≤ 35 y-old

Exclusion Criteria:

* • Wife age > 35 years

  * Frozen semen samples
  * Male partner with severe oligoasthenoteratozoospermia <5 × 106 / mL and 5% progressive motility, included globozoospermia and pinhead samples, and surgically retrieved sperms
  * Poor responder women
  * Women with abnormal endometrium at hCG trigger day.
  * Women with BMI > 31
  * Women with PCOS
  * Previous failed ICSI
  * OHSS)overian hyperstimulation syndrome)
  * Patients with systemic diseases affecting fertility
  * Patients on radiotherapy or receiving medications with gonadotoxic effect eg., chemotherapy

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: prospective cohort study to evaluate seminal plasma lead and cadmium level affects intracytoplasmic sperm injection out come
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The influence of lead and cadmium seminal plasma level on intracytoplasmic sperm injection (ICSI) outcome | baseline
  evaluate the influence of lead (pb) and cadmium (cd) seminal plasma level on embryo development and pregnancy rate during intracytoplasmic sperm injection (ICSI).

REFERENCES:
- [Background] Bernard A. Cadmium & its adverse effects on human health. Indian J Med Res. 2008 Oct;128(4):557-64. PMID 19106447
- [Background] Gill K, Rosiak A, Gaczarzewicz D, Jakubik J, Kurzawa R, Kazienko A, Rymaszewska A, Laszczynska M, Grochans E, Piasecka M. The effect of human sperm chromatin maturity on ICSI outcomes. Hum Cell. 2018 Jul;31(3):220-231. doi: 10.1007/s13577-018-0203-4. Epub 2018 Mar 29. PMID 29594950
- [Background] Wdowiak A, Wdowiak E, Bojar I. Evaluation of trace metals in follicular fluid in ICSI-treated patients. Ann Agric Environ Med. 2017 Jun 23;25(2):213-218. doi: 10.26444/aaem/75422. Epub 2017 Jun 23. PMID 29936824
- [Background] Kumar S, Mishra VV. Review: Toxicants in reproductive fluid and in vitro fertilization (IVF) outcome. Toxicol Ind Health. 2010 Sep;26(8):505-11. doi: 10.1177/0748233710373081. Epub 2010 Jun 7. PMID 20529961
- [Background] Kruger TF, Menkveld R, Stander FS, Lombard CJ, Van der Merwe JP, van Zyl JA, Smith K. Sperm morphologic features as a prognostic factor in in vitro fertilization. Fertil Steril. 1986 Dec;46(6):1118-23. doi: 10.1016/s0015-0282(16)49891-2. PMID 2946611
- [Background] Tong S, Von Schirnding YE, Prapamontol T. [Environmental lead exposure: a public health problem with global dimensions]. Servir. 2000 Jan-Feb;49(1):35-43. No abstract available. Portuguese. PMID 12029976